CLINICAL TRIAL: NCT06512025
Title: Adaptation and Implementation of a Psychoeducational Intervention to Prevent Postpartum Depression and Anxiety Disorders in New Mothers
Brief Title: Implementation of a Psychoeducational Intervention in New Mothers
Acronym: EQEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alba Roca (Other)
Collaborators: Fundació La Marató de TV3 (Other); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor-Investigator, Alba Roca, Doctor, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 193/C/2022
Record Dates: First submitted 2024-07-15; First posted 2024-07-22 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Depression, Postpartum; Anxiety
Keywords: Postpartum Period; Prevention; Preventive Health Care; Psychoeducation; Primiparity; Female
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A CONSORT-compliant parallel group randomized controlled trial will be conducted
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Participants will received the postpartum usual care at the Sexual and Reproductive Health Service (ASSIR).
- WWWT psychoeducative intervention (Experimental): Participants will received the postpartum routine usual care plus two psychoeducative intervention WWWT sessions at the Sexual and Reproductive Health Service (ASSIR).
  Interventions: Behavioral: WWWT psychoeducative intervention

INTERVENTIONS:
Behavioral: WWWT psychoeducative intervention — "What Were We Thinking" (WWWT) is a highly structured, interactive, gender-informed, couples-based, psycho-educational program for parents and a first newborn to promote confident parental caretaking, optimize functioning in the intimate partner relationship and improve infant care manageability.
  The adaptation of the WWWT programme (Catalan and Spanish version) comprises 2 sessions, each lasting 2 hours, that will be designed for groups of 5-7 families - within the first 6 weeks postpartum -, each consisting of mother, partner (or other caregiver) and their infant(s).
  Arms: WWWT psychoeducative intervention

SUMMARY:
The goal of this clinical trial is to implement and examine the clinical effectiveness in a randomized study of the Catalan and Spanish versions of the culturally adapted "What Were We Thinking (WWWT)" psychoeducational intervention in primary care services, with the aim of preventing and reducing the prevalence of postpartum mental illness in new mothers. Additionally, the trial will assess the acceptability and accessibility of the intervention by families and professionals.

Researchers will compare "Usual Care" (standard postnatal care provided by professionals from the Sexual and Reproductive Health Service) with "Intervention group" (usual care plus two psychoeducative intervention WWWT sessions) to see if the "WWWT intervention" is better than "Usual Care" at preventing postpartum depression and anxiety disorders in new mothers.

Participants will:

* Take baseline questionnaires at 2-4 weeks postpartum
* Take usual care or usual care plus two psychoeducative intervention WWWT sessions within the first 6 weeks postpartum
* Take the same questionnaires used in baseline plus a semi-structured interview to diagnose major mental disorder (all participants) at 3 and 6 months follow-up
* Take a brief anonymous self-report survey (only those participants taking the WWWT intervention)

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women
* Given birth a healthy, full-term baby in the preceding 2 weeks
* Receiving postpartum healthcare at Atenció a la salut sexual i reproductiva (ASSIR) of Àrea Integral de Salut Barcelona Esquerra (AIS-BE)
* Over 18 years of age
* Give consent to participate in the study

Exclusion Criteria:

* If are unable to complete the questionnaires due to language or literacy barriers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Mental Disorders | 3 and 6 months postpartum (follow-up)
  The Mini-International Neuropsychiatric Interview (MINI) is a brief structured interview designed for the detection and diagnostic guidance of major Axis I psychiatric disorders as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) and the International Classification of Diseases, 10th Edition (ICD-10). It has an administration time of approximately 15 minutes and is divided into 16 modules, identified by letters, each corresponding to a diagnostic category.
Depressive symptoms | Baseline, 3 and 6 months follow-up
  The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report questionnaire that is used as a screening instrument and for research purposes. Item scores are summed up to a total score (from 0 to 30 points), with higher scores indicating a higher depressive symptom burden. At a cutoff value of 11 (EPDS ≥ 11), the sensitivity of detecting a clinically significant depression is 0.79, the specificity is 0.95, and the positive predictive value is 0.63. The scale has a good internal consistency (Cronbach's α = 0.81).
Depressive symptoms | Baseline, 3 and 6 months follow-up
  The Beck Depression Inventory (BDI-II) is a 21-item self-report instrument designed to assess the severity of depressive symptomatology. In each item, the person evaluated must select the phrase that best describes their condition over the past two weeks from a list of four options, with seven alternatives in items 16 and 18. Each item is scored from 0 to 3 points, with the total score ranging from 0 to 63, with higher scores indicating a higher depressive symptom burden.
Anxiety symptoms | Baseline, 3 and 6 months follow-up
  The Generalised Anxiety Disorder Screener (GAD-7) is a 7-item self-report scale used as a screening instrument measuring symptoms of generalized anxiety disorder that has been recommended as brief screening measure for perinatal anxiety. Item scores are summed up to a total score (from 0 to 21 points), with higher scores indicating a higher anxiety symptom burden. There are no cut-off points established for the Spanish version. In the original version, the authors propose a cut-off point of greater than or equal to 10. For the Spanish version, a Cronbach's alpha coefficient of 0.93 was obtained. Considering the 10-point cutoff, sensitivity values of 86.8% and specificity of 93.4% were found.

SECONDARY OUTCOMES:
Maternal postpartum bonding | Baseline, 3 and 6 months follow-up
  The Postpartum Bonding Questionnaire (PBQ) is a 25-item self-report questionnaire used to evaluate the alterations of the maternal-filial bond in the postpartum period. It includes 4 subscales, with a total of 25 items, which are rated by the mother on a Likert-type scale from 0 to 5. The subscales are general factor, rejection and pathological anger, infant-centered anxiety, and incipient maltreatment scale. The Spanish adaptation and validation has an adequate psychometrics property for use with clinical and general population of Spanish puerperal women. The PBQ could be summarized in a general factor and that the use of the total score of the scale would already be useful to detect alterations in the mother-infant bond (Cronbach's alpha reliability value of 0.90). A total score of 26 or more would indicate some type of attachment disorder, and a score of 40 or more would indicate the presence of maternal rejection or a severe attachment disorder.
Parenting self-regulation | Baseline, 3 and 6 months follow-up
  The Me as a Parent scale (MaaPs) is a 16-item self-report scale used to measure the parents' perceptions of their parenting role. The scale has four theoretical sub-dimensions (Parenting Self-Efficacy; Personal Agency; Self-Management; and Self-Sufficiency), each containing four items scored on a 5-point agreement scale, with a total scale score range of 16-80. Higher scores indicate a higher parent's self-perceived competence and efficacy.
Marital Adjustment | Baseline, 3 and 6 months follow-up
  The Escala de Ajuste Diádico (EAD-13) is a 13-item self-report short version of the Dyadic Adjustment Scale (DAS) used to assess the degree of harmony or adjustment between the members of the couple's relationship through 3 dimensions: consensus (capacity, resources and skills to reach agreements or find joint solutions to problems), satisfaction (level of well-being, happiness and commitment in the couple) and cohesion (degree of involvement of one member of the couple with the other). Item scores are summed up to a total score (from 12 to 75 points), with higher scores indicating increased marital adjustment. The scale has shown adequate psychometric properties to be applied in the Spanish context, finding a Cronbach's alpha reliability value of 0.81.
Satisfaction survey | Intervention group participants immediately after completing the WWWT psychoeducative group.
  Satisfaction survey is made up of Likert-type questions from 0 to 5 points
  (1 = completely disagree, 5 = completely agree) and open questions to measure participants' satisfaction with the WWWT psychoeducational intervention in terms of accessibility, comprehensibility, acceptability and usefulness, and identify needs or possible difficulties in its implementation.

OTHER OUTCOMES:
Partner Violence | Baseline, 3 and 6 months follow-up
  The Woman Abuse Screening Tool (WAST) is 8-item self-report screening instrument for intimate partner physical, emotional and/or sexual violence. The items are answered on a scale of intensity or frequency of 3 degrees. The maximum score range of the scale ranges from 8 to 24, which is obtained from the sum of the responses of the 8 items of the scale. Higher scores indicate a higher risk of partner abuse. The scale It was translated and validated in Spanish population and finding good internal consistency (Cronbach's α = 0.95).
Alcohol use | Baseline, 3 and 6 months follow-up
  The Alcohol Use Disorders Identification Test (AUDIT-C) is a shortened version of the AUDIT, comprising the initial three items. It is designed to facilitate the expedient identification of individuals engaging in hazardous alcohol consumption. Total scores range from 0 to 12, with elevated scores indicating heightened risk-taking drinking behaviors. The sensitivity of the AUDIT-C has been demonstrated to range from 54 to 98%, while its specificity has been shown to range from 57 to 93%, depending on the definition of heavy drinking employed
Childhood trauma | Baseline
  The Early Trauma Inventory Self Report Short-Form (ETISR-SF) is a 27-item self-report inventory that retrospectively assesses the presence of traumatic events experienced before and after the age of 18. It contains dichotomous items (yes or not) that assess general trauma, emotional, physical, or sexual abuse. The ETI-SF internal consistency ranged between 0.42 and 0.72, and test-retest reliability ranged from 0.84 to 0.96.
Vulnerable Personality Style | Baseline
  The Vulnerable Personality Style Questionnaire (VPSQ) is a 9-item self-report scale used to assess personality traits which increase the risk of postpartum depression (coping, nervy, timidity, sensitivity, worrier, organised, obsessive, expressive and volatility). It is rated on a 5-point Likert scale (1 = "not at all" to 5 = "very much so"). Total scores range from 9 to 45, and higher scores indicate increased vulnerability.
Perceived Social Support | Baseline, 3 and 6 months follow-up
  The Multidimensional Perceived Social Support Scale (MSPPSS) is a 12-item measure of perceived adequacy of social support from three sources: family, friends and significant other; using a 5-point Likert scale (0 = strongly disagree, 5 = strongly agree).
Sociodemographic variables | Baseline
  Age, country of birth, current marital status, occupation prior to having the infant, highest level of education completed, employment, will be collected by an ad hoc questionnaire.
Psychiatric history, clinical and health variables | Baseline
  Self-rated general health, maternal rating of infant general health, history of diagnosed mental health problems (included substance use) and history of physical and sexual abuse will be collected by an Ad hoc questionnaire.
Obstetrical and neonatal outcomes | Baseline
  Obstetric history (previous pregnancies and abortions), type of conception (spontaneous or using Assisted Reproductive Technology), unplanned pregnancy, mode of birth, singleton infant or multiples, sex of infant, birth weight (grams), week of pregnancy when delivery took place, overall birth experience, and method of feeding the baby (breastfeeding, mixed feeding, bottle feeding) will be assessed by an Ad hoc questionnaire.
Baby's temperament | Baseline, 3 and 6 months follow-up
  The Baby Temperament Scale is a 10-item scale that allows obtaining an individualized profile of 9 basic temperamental traits, and a classification between three pure categories: slow child, difficult child and active child. Each dimension allows three response options: two opposite and one intermediate. It is not an instrument with psychometric validation.

CONTACTS AND LOCATIONS:
Overall Officials: Alba Roca, Doctor, Principal Investigator — Fundacion Clinic per a la Recerca Biomédica
Locations (2):
- Spain (2):
  - Unitat de Salut Mental Perinatal (USMP) de l'Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Atenció a la salut sexual i reproductiva (ASSIR) de l'Àrea Integral de Salut Barcelona Esquerra (AIS-BE), Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No